CLINICAL TRIAL: NCT05573438
Title: Acute Inflammatory and Metabolic Effect of High Fructose Intake in Normal Weight Women: Double Blind, Randomized Crossover Study.
Brief Title: Acute Inflammatory and Metabolic Effect of High Fructose Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adaliene Versiani M. Ferreira (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Adaliene Versiani M. Ferreira, Clinical Professor, Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CAAE: 21852314.7.0000.5149
Record Dates: First submitted 2022-09-22; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Inflammatory Response; Metabolic Disturbance
Keywords: Fructose; Postprandial Period; Inflammation; Metabolism
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: This will be a three-arm crossover, randomized, double-blind clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fructose (Experimental): Participants received a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with fructose. The meals provided 25% of the energy requirements. The meal consisted of 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of fructose).
  Interventions: Other: Group fructose
- Sucrose (Experimental): Participants received a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with sucrose. The meals provided 25% of the energy requirements. The meal consisted of 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of sucrose).
  Interventions: Other: Group Sucrose
- Glucose (Placebo Comparator): Participants received a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with glucose. The meals provided 25% of the energy requirements. The meal consisted of 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of glucose).
  Interventions: Other: Group Glucose

INTERVENTIONS:
Other: Group fructose — Participants will receive a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with fructose. The meals will provide 25% of the energy requirements, calculated from the resting energy expenditure measured by indirect calorimetry (KORR®, MetaCheck) multiplied by the activity factor (24) plus 10% referring to the thermal effect of food. The meal will have 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of fructose. The sweetened drinks will have artificial fruit flavor to avoid the identification of the content by the researchers and the volunteers.
  Arms: Fructose
Other: Group Sucrose — Participants will receive a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with sucrose. The meals will provide 25% of the energy requirements, calculated from the resting energy expenditure measured by indirect calorimetry (KORR®, MetaCheck) multiplied by the activity factor (24) plus 10% referring to the thermal effect of food. The meal will have 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of sucrose. The sweetened drinks will have artificial fruit flavor to avoid the identification of the content by the researchers and the volunteers.
  Arms: Sucrose
Other: Group Glucose — Participants will receive a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with glucose. The meals will provide 25% of the energy requirements, calculated from the resting energy expenditure measured by indirect calorimetry (KORR®, MetaCheck) multiplied by the activity factor (24) plus 10% referring to the thermal effect of food. The meal will have 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of glucose. The sweetened drinks will have artificial fruit flavor to avoid the identification of the content by the researchers and the volunteers.
  Other Names: Placebo Comparator
  Arms: Glucose

SUMMARY:
Fructose consumption is associated with the development of metabolic diseases and low-grade inflammation. However, the acute effect of a single meal rich in fructose on the metabolic and inflammatory response is not fully understood. This study will to evaluate the acute metabolic and inflammatory effect caused by a meal containing fructose overload. This will be a three-arm crossover, randomized, double-blind clinical trial.

Participants will undergo the three interventions for random order: (i) standardized meal plus sucrose overload; (ii) standardized meal plus glucose overload; (iii) standardized meal plus fructose overload. During the washout period (7 to 21 days), the subjects will instructed to maintain their usual eating behavior and physical activity.

On the day of each intervention, participants will to the outpatient clinic in the morning after an overnight fast. Anthropometric data (weight, height, and waist circumference) will collected. Body composition will evaluated using bioimpedance (Quantum® apparatus, RJM Systems, Michigan) and blood pressure and heart rate (digital monitor, model HEM705CP®, Omron) will measured after 30 minutes of rest.

A catheter with a three-way stopcock will inserted into the arm of the volunteers. Blood samples (5mL) will collected after overnight fasting (baseline) and 30, 60, 120, and 240 minutes after the standardized meal containing sucrose or glucose or fructose overload. Participants will remain seated throughout the evaluation period. Participants will receive a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with similar amounts of different carbohydrates (sucrose, glucose, or fructose) in each intervention. The meals will provide 25% of the energy requirements, calculated from the resting energy expenditure measured by indirect calorimetry (KORR®, MetaCheck) multiplied by the activity factor plus 10% referring to the thermal effect of food. The meal will consiste of 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of sucrose or glucose or fructose).

Serum levels of glucose, triglycerides, total cholesterol, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) will be measured by colorimetric enzymatic test. Serum levels of adiponectin, leptin, resistin and TNF will be measured by Enzyme Linked ImmuneSorbent Assay (ELISA). Serum levels of IL-2, IL-4, IL-5, IL-6, IL-10, IL-17, IFN-γ and eotaxin will be obtained by the Cytometric Bead Array (CBA).

DETAILED DESCRIPTION:
This will be a three-arm crossover, randomized, double-blind clinical trial performed at the Alpha Institute of Gastroenterology of the Hospital das Clínicas (Belo Horizonte, MG, Brazil). All experimental procedures will be conducted according to the guidelines laid down in the Declaration of Helsinki. The research protocol was approved by the Institutional Review Board of the Universidade Federal de Minas Gerais (CAAE: 21852314.7.0000.5149). All volunteers will signed the informed consent prior to the start of the study.

Sample The sample size of 17 subjects was calculated considering the minimum number of participants to detect a difference of at least 11 mg/dL in the levels of triglycerides, 1.2 ng/mL in adiponectin and 1.9 pg/mL in TNF (pilot study) before and after the intake of a single meal containing a fructose overload, 95% confidence interval and statistical power of the 80%.

Study design Each participant will in three visits with washout period between 7 and 21 days. At each visit, the participant will pass by a different intervention. Three interventions will curr in random order: (i) standardized meal plus sucrose overload; (ii) standardized meal plus glucose overload; (iii) standardized meal plus fructose overload. During the washout period, the subjects will instructed to maintain their usual eating behavior and physical activity. Participants will instructed to avoid consuming caffeine and alcoholic beverages and perform intense physical activity within 24 hours before each visit.

On the day of each intervention, participants will go to the outpatient clinic in the morning after an overnight fast. Anthropometric data (weight, height, and waist circumference) will collected. Body composition will evaluated using bioimpedance (Quantum® apparatus, RJM Systems, Michigan) and blood pressure and heart rate (digital monitor, model HEM705CP®, Omron) will measured after 30 minutes of rest.

A catheter with a three-way stopcock will inserted into the arm of the volunteers. Blood samples (5mL) will collected after overnight fasting (baseline) and 30, 60, 120, and 240 minutes after the standardized meal containing sucrose or glucose or fructose overload. Participants remained seated throughout the evaluation period.

Intervention Participants will receive a standardized meal of bread, ham, and margarine plus a sweetened drink (200mL) with similar amounts of different carbohydrates (sucrose, glucose, or fructose) in each intervention. The meals will provide 25% of the energy requirements, calculated from the resting energy expenditure measured by indirect calorimetry (KORR®, MetaCheck) multiplied by the activity factor plus 10% referring to the thermal effect of food. The meal will consiste of 15% of protein, 30% of fat, and 55% of carbohydrate (30% of complex carbohydrates and 25% of sucrose or glucose or fructose). The sweetened drinks will have artificial fruit flavor to avoid the identification of the content by the researchers and the volunteers.

The amount of refined offered carbohydrates to the participants (18 - 25g in a single meal) will considered an overload since the World Health Organization and the National Center for Chronic Disease Prevention and Health Promotion recommend that the consumption of added sugars should not exceed 10% of the total daily calories. For example, in a 2.000 caloric diet, no more than 200 calories should come from added sugars (about 12 teaspoons). In addition, several authors who investigated short- and long-term (≥ 3 weeks) fructose consumption in metabolic and inflammatory biomarkers offered 25% of total energy expenditure (GET) in the form of sucrose, glucose, fructose or high fructose corn syrup per day. On the other hand, the amount of these carbohydrates offered in the present study is part of the eating routine of many individuals (e.g., 200mL of regular soda contains 21 grams of sucrose).

Blood analysis Serum levels of glucose, triglycerides, total cholesterol, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) will measured by colorimetric enzymatic test (Bioclin®, Belo Horizonte, MG, Brazil). Serum levels of adiponectin, leptin, resistin and TNF will measured by Enzyme Linked ImmuneSorbent Assay (ELISA) following the manufacturer's instructions (R&D Systems®). Serum levels of IL-2, IL-4, IL-5, IL-6, IL-10, IL-17, IFN-γ and eotaxin will obtained by the Cytometric Bead Array (CBA) method (BD Bioscience, San Diego, CA, USA) in flow cytometry. Collected blood will diluted in Turk's solution. The number of total white blood cell will obtained using a Neubauer chamber (×40 objective).

Statistical Analyses All quantitative variables will present as mean ± standard error (SEM). The normality of the quantitative variables will tested through the Shapiro-Wilk test. Student's t Simple and Mann-Whitney tests will allow comparisons between the initial characteristics of those who completed the study and those who did not, and between volunteers who will participate in the sub-sample and those who not. To compare the anthropometric and clinical characteristics between baseline and the subsequent assessments, we will use the ANOVA test for repeated measures 1-factor or Kruskal-Wallis according to the normality followed by Bonferroni post-test. Postprandial metabolic and inflammatory markers will compared by the Generalized Equation of Estimates (GEE) model to evaluate the effect of group allocation (carbohydrate type), time and adjusting for time-group effect (interaction). The variables will treated with the connection range function and the correlation matrix will the covariance of an unstructured and robust estimator. The Bonferroni post-test will identifie the presence of signifcant effects. Significance will set at P < 0.05. The data will analysed using the Statistical Package for the Social Sciences (SPSS) software version 20 and GraphPad Prism version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Women aged
* 20 and 47 years
* body mass index (BMI) from 18.50 to 24.99 kg/m²

Exclusion Criteria:

* chronic diseases, such as DM, chronic renal failure (CRF), cardiovascular or hepatic diseases, acute inflammatory or autoimmune diseases;
* participants with glycemia > 99 mg/dL;
* triglycerides > 200 mg/dL;
* prior bariatric surgery for weight loss;
* people who were taking medication for thyroid disorders, dyslipidemia, insulin sensitivity or DM, CRF, cardiovascular and hepatic diseases, inflammation and/or infection, immunosuppressive and weight loss;
* smokers or people who drink more than two doses of alcohol a day (28g of pure alcohol); and (vii) pregnancy or breast-feeding.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in serum levels of triglycerides | Change from Baseline serum level at 240 minutes postprandial.
  Triglycerides (ml/dL)
Changes in serum levels of adiponectin | Change from Baseline serum level at 240 minutes postprandial.
  Adiponectin (pg/dL)
Changes in serum levels of tumor necrosis factor | Change from Baseline serum level at 240 minutes postprandial.
  Tumor necrosis factor (pg/dL)

SECONDARY OUTCOMES:
Changes in serum levels of interleukin-2 | Change from Baseline serum level at 240 minutes postprandial.
  Interleukin-2 (pg/dL)
Changes in serum levels of interleukin-4 | Change from Baseline serum level at 240 minutes postprandial.
  Interleukin-4 (pg/dL)
Changes in serum levels of interleukin-5 | Change from Baseline serum level at 240 minutes postprandial.
  Interleukin-5 (pg/dL)
Changes in serum levels of interleukin-6 | Change from Baseline serum level at 240 minutes postprandial.
  Interleukin-6 (pg/dL)
Changes in serum levels of interleukin-10 | Change from Baseline serum level at 240 minutes postprandial.
  Interleukin-10 (pg/dL)
Changes in serum levels of interleukin-17 | Change from Baseline serum level at 240 minutes postprandial.
  Interleukin-17 (pg/dL)
Changes in serum levels of interferon gamma | Change from Baseline serum level at 240 minutes postprandial.
  Interferon gamma (pg/dL)
Changes in serum levels of ofeotaxin | Change from Baseline serum level at 240 minutes postprandial.
  Ofeotaxin (pg/dL)
Changes in serum levels of glucose | Change from Baseline serum level at 240 minutes postprandial.
  Glucose (mg/dL)
Changes in serum levels of cholesterol | Change from Baseline serum level at 240 minutes postprandial.
  Cholesterol (mg/dL)
Changes in serum levels of Aspartate aminotransferase | Change from Baseline serum level at 240 minutes postprandial.
  Aspartate aminotransferase (U/L)
Changes in serum levels of Alanine aminotransferase | Change from Baseline serum level at 240 minutes postprandial.
  Aspartate aminotransferase (U/L)
Changes in serum levels of Leptin | Change from Baseline serum level at 240 minutes postprandial.
  Leptin (pg/dL)
Change in metabolic profile | Change from Baseline serum level at 240 minutes postprandial.
  Resistin (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Adaliene VM Ferreira, PhD, Principal Investigator — Federal University of Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigues AMDS, Martins LB, Fagundes GBP, Tibaes JRB, Amaral MHA, Vieira ELM, Oliveira MC, Correia MITD, Ferreira AVM. Acute inflammatory and metabolic effect of high fructose intake in normal-weight women: A randomized, double-masked, crossover trial. Nutrition. 2025 Jan;129:112602. doi: 10.1016/j.nut.2024.112602. Epub 2024 Oct 9. PMID 39442382